CLINICAL TRIAL: NCT01250015
Title: THE RESULTS OF A RANDOMISED CONTROLLED QUESTIONNAIRE-BASED TRIAL ON WHETHER PROVISION OF NUMERICAL AND PICTORIAL INFORMATION ON RISK AND BENEFIT AFFECTS THE UPTAKE OF COLORECTAL CANCER SCREENING?
Brief Title: Does Numerical And Pictorial Information On Risk And Benefit Affects The Uptake Of Colorectal Cancer Screening?
Status: Completed | Type: Observational
Sponsor: County Durham and Darlington NHS Foundation Trust (Other Government)
Collaborators: Internal funding Local Gastroenterology Research fund (Questionnaire only study) (Unknown)
Responsible Party: Peter Trewby, county darlington and durham NHS foundation trust
Other Study IDs: 1; CDDFT (UK) (Other: CDDFT, UK); CDDFT, UK (Other: CDDFT, UK)
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2008-03

CONDITIONS: Colorectal Cancer Screening
Keywords: colorectal cancer; consent; screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- control: given standard nhs advice leaflet
- interventional: given standard nhs advice leaflet with numerical information and pictograms

SUMMARY:
To establish whether provision of numerical data, framed as event rates and illustrated by pictograms, and including figures for all-cause mortality, affects subjects' attitudes to colorectal cancer (CRC) screening.

Design and Intervention. Randomised questionnaire and telephone study comparing the responses of a control group given the standard National Health Service (NHS) CRC screening information with the responses of an intervention group given the same information but enhanced with additional numerical and pictorial information.

Setting

ELIGIBILITY:
Inclusion Criteria:

Age 60 - 70

-

Exclusion Criteria:

* No previous cancer or previous colonoscopy Not able to give informed consent

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects attending GP and hospital outpatients
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Comparison of the two groups' overall wish to be screened | 1 year
  The study compared the two groups' overall wish to be screened as recorded by questionnaire

SECONDARY OUTCOMES:
Impact of different summary points on subject's desire to be screened | 1 year
  The impact of each of the 6 summary points in the NHS information leaflet on the subject's desire to be screened depending on whether or not they were enhanced by numerical and pictorial information, the summary point that most influenced their decision on whether to be screened; and the views of the intervention group on the numerical and pictorial information provided

CONTACTS AND LOCATIONS:
Locations (1):
- Darlington Memorial Hospital, Darlington, Co Durham, United Kingdom

REFERENCES:
- See also: CDDFT, NHS, UK — http://www.nhs.uk/Services/Hospitals/Overview/DefaultView.aspx?id=2241